CLINICAL TRIAL: NCT01234480
Title: Intended Use Study of the BD SurePath Plus™ Pap
Status: Terminated | Type: Interventional
Why Stopped: Decided not to pursue commercialization of the product
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TPO-10-06084
Record Dates: First submitted 2010-10-14; First posted 2010-11-04 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Uterine Cervical Neoplasms; Uterine Cervical Cancer; Neoplasms, Squamous Cell; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Papilloma
Keywords: Liquid based cytology; Surepath
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms, Squamous Cell; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Papilloma | interventions — Papanicolaou Test; Colposcopy; Human Papillomavirus DNA Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Participants with Cervical Disease (Experimental): Participants positive for Cervical Disease (CIN2 or higher) as determined by adjudicated histology from biopsy/ECC.
  Interventions: Device: BD SurePath Plus Pap test; Device: BD SurePath Pap test; Procedure: colposcopy with biopsy/ECC; Device: HPV DNA test
- Participants without Cervical Disease (Experimental): Participants negative for Cervical Disease (CIN2 or higher) as determined by adjudicated histology from biopsy/ECC.
  Interventions: Device: BD SurePath Plus Pap test; Device: BD SurePath Pap test; Device: HPV DNA test

INTERVENTIONS:
Device: BD SurePath Plus Pap test — BD SurePath Plus Pap test
Device: BD SurePath Pap test — BD SurePath Plus Pap test
Procedure: colposcopy with biopsy/ECC — Colposcopy with biopsy/ECC for subjects with 1)BD SurePath Pap NILM, but HPV positive, or 2) BD SurePath Plus Pap test result of ASC-US or higher 3)BD SurePath Pap ASC-US or higher
  Arms: Participants with Cervical Disease
Device: HPV DNA test — digene HC2 HPV DNA test
  Other Names: digene HC2 HPV DNA test

SUMMARY:
This study will provide data on the performance of the BD SurePath Plus™ Pap test for identifying high grade cervical disease. This study will be conducted with approximately 12,500 women undergoing routine cervical cancer screening, of whom women with abnormal cytology and/or positive HPV test will be selected to undergo colposcopy and biopsy/ECC. Subjects with abnormal cytology results with biopsy results of less than or equal to CIN1 or CIN2 untreated will be asked to return in 6-8 months for follow-up testing. Subjects may be asked to proceed to a longer-term follow-up study and undergo cytological evaluation annually for 3 years (separate study).

DETAILED DESCRIPTION:
This is a pivotal, multi-center in vitro diagnostic study comparing the BD SurePath Plus Pap test to current practice (cytologic examination utilizing the BD SurePath liquid-based Pap test with conjunctive HPV testing) for the detection of cervical cancer and high-grade cervical disease (collectively referred to as CIN2+) in women.

The new BD SurePath Plus Pap Test combines a traditional Papanicolaou staining for cellular morphology, with brown nuclear immunostaining resulting from the over-expression of specific protein biomarkers, on one slide, to improve the detection of high-grade cervical disease and cervical cancer (collectively referred to as CIN2+).

ELIGIBILITY:
Inclusion Criteria:

Study subjects must give voluntary written informed consent to participate in this study.

- Females ages 18 - 35 years, inclusive; or women at high- risk for cervical cancer or its precursor lesions.

High-risk is defined as:

* Have had a previous high-risk HPV positive test in the last 5 years; or
* Have had an abnormal Pap test (ASC-US or higher) in the last 5 years; or
* Have not been screened for cervical cancer by either a Pap test or HPV test in the last 5 years.

Exclusion Criteria:

* Subjects who are 36 years of age or greater who are not high risk, and/or:

  1. Have not had an abnormal Pap in the last 5 years; or
  2. Have not had a positive HPV test in the last 5 years; or
  3. Have been screened in the last 5 years without an abnormal Pap or HPV result
* Subjects known to be pregnant or planning to become pregnant prior to the potential six months follow-up visit (self-reported). Subjects who decide to become pregnant prior to the six-month follow up visit or found to be pregnant after the first visit, but prior to the six-month follow-up visit will be terminated from further study participation at that time
* Subjects who have had a prior complete or partial hysterectomy involving removal of the cervix.
* Subjects who have had an application of chemical compounds to the cervical area within the 24 hours prior to study entry, e.g., acetic acid, iodine, spermicide, douche, anti-fungal medications, etc.
* Subjects on whom conization, LEEP, laser surgery, or cryosurgery has been performed within the past five months.
* Subjects currently undergoing radiation and/or chemotherapy.
* Subjects under the age of 18.
* Subjects who have previously received a HPV vaccine with any number of doses.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5859 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Women's: Health, Research, Gynecology, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All Enrolled Participants - Cervical cancer status was not known upon enrollment
Period: Overall Study
Arm/Group | All Study Participants
Started | 5859
Completed | 5416
Not Completed | 443
Not completed — Pregnancy | 88
Not completed — >36/Normal History | 50
Not completed — Age | 3
Not completed — HPV Vaccine History | 28
Not completed — HPV Vaccine after Enrollment | 17
Not completed — Hysterectomy | 2
Not completed — Hysterectomy post enrollment | 1
Not completed — Inclusion/Exclusion Violation | 3
Not completed — Informed Consent Form Violation | 30
Not completed — Incorrect Visit | 3
Not completed — No Florida Lab License | 20
Not completed — Out of Window | 42
Not completed — Sample Processing/Storage | 92
Not completed — Site Amendment prohibited colposcopy | 11
Not completed — Site/Subject non-compliance | 44
Not completed — Missing Sample | 9

BASELINE CHARACTERISTICS:
Population: Participants with evaluable samples.
Groups:
- All Evaluable Participants: All participants with satisfactory samples at completion of the study.
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 3731
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3731
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3731
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 889
  Not Hispanic or Latino | 2842
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3731

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity, Specificity, PPV, and NPV of BD SurePath Plus Pap Test for the Determination of Cervical Disease as Defined by CIN2 or Higher
Description: Estimate the sensitivity, specificity, positive predictive value and negative predictive value of the BD SurePath Plus Pap test in detecting cervical disease as defined as CIN2 or higher
Time Frame: 10 months
Population: All evaluable non-missing samples.
Measure: Number (95% Confidence Interval); unit: Percent
Groups:
- SurePath Plus: Samples tested on the SurePath Plus
- SurePath Pap: Samples tested on the SurePath Pap
Arm/Group | SurePath Plus | SurePath Pap
Number analyzed (Participants) | 3731 | 3731
Percent
  Sensitivity (ASC-US+) | 84.9 [77.4 to 90.2] | 71.4 [62.7 to 78.8]
  Specificity (ASC-US+) | 84.7 [83.5 to 85.9] | 88.7 [87.5 to 89.7]
  PPV (ASC-US+) | 16.7 [15.1 to 18.2] | 18.5 [16.2 to 20.7]
  NPV (ASC-US+) | 99.4 [99.0 to 99.6] | 98.9 [98.5 to 99.1]
  Sensitivity (ASC-H+) | 65.5 [56.6 to 73.5] | 43.7 [35.1 to 52.7]
  Specificity (ASC-H+) | 92.2 [91.2 to 93.1] | 94.4 [93.5 to 95.1]
  PPV (ASC-H+) | 23.2 [20.1 to 26.3] | 21.8 [17.8 to 26.1]
  NPV (ASC-H+) | 98.7 [98.3 to 99.0] | 97.9 [97.6 to 98.2]
  Sensitivity (LSIL+) | 58.0 [49.0 to 66.5] | 40.3 [32.0 to 49.3]
  Specificity (LSIL+) | 93.4 [92.5 to 94.2] | 94.7 [93.8 to 95.4]
  PPV (LSIL+) | 24.0 [20.4 to 27.6] | 21.4 [17.2 to 25.9]
  NPV (LSIL+) | 98.4 [98.1 to 98.7] | 97.8 [97.5 to 98.1]
  Sensitivity (HSIL+) | 37.8 [29.6 to 46.8] | 16.0 [10.5 to 23.6]
  Specificity (HSIL+) | 98.3 [97.8 to 98.7] | 99.8 [99.6 to 99.9]
  PPV (HSIL+) | 45.0 [36.5 to 53.3] | 76.0 [56.9 to 88.3]
  NPV (HSIL+) | 97.8 [97.5 to 98.1] | 97.1 [96.9 to 97.3]

2. Secondary Outcome: Compare the Sensitivity and Specificity of the BD SurePath Plus Pap Test to the SurePath Pap With HPV Reflex Testing for CIN2+ Disease Detection.
Time Frame: 10 months
Population: Evaluable samples that had also had HPV reflex testing
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- SurePath Plus With Immunostain: Samples tested on the SurePath Plus
- SurePath Pap With HPV: Samples tested on the SurePath Pap
Arm/Group | SurePath Plus With Immunostain | SurePath Pap With HPV
Number analyzed (Participants) | 221 | 221
percent
  Sensitivity (ASC-US) | 78.8 [62.2 to 89.3] | 87.9 [72.7 to 92.5]
  Specificity (ASC-US) | 45.7 [38.8 to 52.9] | 41.5 [34.7 to 48.6]

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | All Evaluable Participants
All-Cause Mortality (participants affected / at risk) | 0/3731
Serious Adverse Events (participants affected / at risk) | 0/3731
Other Adverse Events (participants affected / at risk) | 0/3731

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No